CLINICAL TRIAL: NCT06361030
Title: An Exploratory Clinical Study of Surufatinib Combined With Gemcitabine Plus Nab-paclitaxel in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Surufatinib Combined With Gemcitabine Plus Nab-paclitaxel in Locally Advanced Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-C2-PC01
Record Dates: First submitted 2024-04-01; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer; Pancreatic Cancer Non-resectable; Pancreatic Ductal Adenocarcinoma, PDAC
Keywords: Pancreatic ductal adenocarcinoma; surufatinib; surgical conversion; gemcitabine; nab-paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms; Anophthalmia with pulmonary hypoplasia | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): After 4-6 cycles of induction therapy with gemcitabine and nab-paclitaxel plus surufatinib, if become operable, the therapy will be continued for another 6 months after surgery; if not operable, the therapy will be also continued as long as no PD during induction therapy. If PD occurs, it will enter second-line therapy.
  Interventions: Drug: surufatinib combined with gemcitabine plus nab-paclitaxel

INTERVENTIONS:
Drug: surufatinib combined with gemcitabine plus nab-paclitaxel — Surufatinib capsules: oral, once daily. Combination treatment period: 200 mg each time, every 4 weeks for a treatment cycle(Q4W). If all the chemotherapy drugs were stopped during the maintenance treatment period, only surufatinib was left, the dose of Surufatinib could be increased to 300 mg per dose according to the patient's condition.
  Gemcitabine: iv, 1000 mg/m2, days 1, 8, and 15 of each treatment cycle, Q4W. Paclitaxel (albumin-bound), iv, 125mg/m2, on days 1, 8 and 15 of each treatment cycle, Q4W.
  All they will be used until disease progression, death, intolerable toxicity, initiation of new antineoplastic therapy, withdrawal of consent, loss to follow-up, or any other protocol-specified event requiring treatment discontinuation or study closure, whichever occurred first.
  But If surgical resection was performed, they will be only maintained for 6 months after surgery.

SUMMARY:
To evaluate the efficacy and safety of surufatinib combined with gemcitabine plus nab-paclitaxel in patients with locally advance d pancreatic cancer

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) has a very poor prognosis. Currently, there is no standard treatment for locally unresectable PDAC, and clinical research and conversion therapy are encouraged by guidelines. Whether it is conversion or palliative chemotherapy, in fact, the choice of chemotherapy is based on the existing first-line regimens of metastatic PDCA. Gemcitabine combined with nab-paclitaxel is one of the preferred first-line chemotherapy regimens for metastatic or locally advanced PDAC. However, the conversion rate of gemcitabine combined with nab-paclitaxel is not ideal according to the current results. The aim of this study is to investigate whether the combination of gemcitabine and nab-paclitaxel with surufatinib can improve the surgical conversion rate.

This is a prospective, single-arm exploratory clinical study. A safety run-in period of 6 patients will be set. After 4-6 cycles of induction therapy with gemcitabine and nab-paclitaxel plus surufatinib, if become operable, the therapy will be continued for another 6 months after surgery; if not operable, the therapy will be also continued as long as no PD during induction therapy. If PD occurs, it will enter second-line therapy. Surufatinib capsule will be administered orally 200mg, once daily, a 4-week treatment cycle(Q4W) during combined with gemcitabine and nab-paclitaxel. If all chemotherapy drugs are stopped during the maintenance treatment period and only surufatinib is left, the dose of surufatinib can be increased to 300 mg per dose according to the patient's condition. Gemcitabine and nab-paclitaxel plus surufatinib will be used until disease progression, death, intolerable toxicity, initiation of new antineoplastic therapy, withdrawal of informed consent, loss of follow-up, and other conditions that require treatment discontinuation or the study is completed. Whichever comes first. If surgical resection was performed, it will be maintained for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study and signed the informed consent, with good compliance and follow-up;
2. Aged 18-75 years old (including 18 and 75 years old)
3. male or female
4. Histologically or cytologically confirmed adenocarcinoma of the pancreas
5. Unresectable pancreatic cancer according to radiographic criteria (CT or MRI scans) or exploration( NCCN guidelines were referred): (1)The portal and superior mesenteric vein could not be reconstructed safely due to tumor invasion, venous occlusion, or involvement of a large area of the superior mesenteric vein jejunal branch (2)If pancreatic head/uncinate tumor: tumor contacts superior mesenteric artery or celiac trunk artery >180 degrees. If pancreatic body tail tumor: tumor contacts the superior mesenteric artery or celiac trunk artery>180 degrees, and tumor contacts the celiac trunk artery and infiltrates the abdominal aorta.
6. Without distant metastasis as defined by CT or MRI scan of the chest, abdomen and pelvis
7. No prior systematic treatment for advanced pancreatic cancer
8. At least one measurable lesion was required. (Response evaluation criteria in Solid Tumors, RECIST, version 1.1)
9. ECOG performance status of 0 or 1
10. Expected survival ≥12 weeks
11. Acceptable organ and bone marrow function, laboratory values within 7 days prior to enrollment (no blood components, cell growth factors, albumin, or other corrective medications were allowed within 14 days prior to laboratory testing), as follows: (1)Blood routine: neutrophils ≥ 1.5 x 10⁹/L, platelets ≥ 100 x 10⁹/L, hemoglobin ≥ 9.0g/dL; (2) Liver function: serum total bilirubin ≤ 1.5 x ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤2.5 × ULN in subjects without liver metastases, AST and ALT levels ≤5 × ULN in subjects with documented liver metastases; (3) Renal function: serum creatinine ≤ 1.5 x ULN, or creatinine clearance (CCr) ≥ 50mL/min; Urine protein < 2 +; if urine protein ≥2+ at baseline, 24-hour urine collection should be done and 24-hour urine protein < 1g; (4) Coagulation function: international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN.
12. Female subjects of childbearing potential or male subjects whose sexual partner is a female of childbearing age should take effective contraceptive measures during the whole treatment period and 6 months after the last treatment.

Exclusion Criteria:

1. Participants had a second primary malignancy detected prior to the first dose of study treatment, or has other malignancies diagnosed within 5 years prior to the first dose of study treatment, with the exception of radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radically resected carcinoma in situ;
2. Allergy to study medication or excipients
3. With dysphagia or known malabsorption of drugs
4. Have participated in any other drug clinical trial and received the corresponding trial drug within the previous 4 weeks. Or are participating in other clinical studies that may interfere with this study.
5. Drug-uncontrolled hypertension；systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg; History of hypertensive crisis or hypertensive encephalopathy.
6. Patients with active gastric or duodenal ulcer, ulcerative colitis, intestinal obstruction, other gastrointestinal diseases, or active bleeding from unresectable tumors before enrollment, or other conditions that may cause gastrointestinal bleeding or perforation as judged by the investigator; Or have a history of bowel perforation or fistula and do not fully recover from surgery.
7. Patients had a history of arterial or deep-vein thrombosis within 6 months before enrollment ，or had evidence or history of bleeding tendency, regardless of severity, within 2 months before enrollment.
8. Stroke or transient ischemic attack occurred within 12 months before enrollment.
9. Incomplete healing of skin wounds, surgical sites, trauma sites, severe mucosal ulcers, or fractures.
10. Active bacterial, viral, or fungal infections requiring systemic treatment, defined as signs/symptoms associated with the infection that persist and do not improve despite appropriate antibiotic, antiviral, and/or other treatments
11. Known hepatitis B or C infection or a history of human immunodeficiency virus (HIV) infection ; Subjects receiving immunosuppressive or myelosuppressive drugs is considered to be associated with an increased risk of severe neutropenia complications by the investigators.
12. Severe cardiovascular disease, including unstable angina or myocardial infarction, occurred within 6 months before enrollment; Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting within 6 months before enrollment; New York Heart Association (NYHA) classification of congestive heart failure >Grade 2; Ventricular arrhythmias requiring medical therapy; LVEF(left ventricular ejection fraction)<50%. Electrocardiogram (ECG) corrected QT interval ≥480 msec.
13. Clinically significant ascites
14. Clinically significant electrolyte disturbances.
15. Severe mental illness that may compromise the safety of the subjects or the integrity of the study data.
16. Any clinical or laboratory abnormalities or adherence that were deemed by the investigator to be inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Surgical conversion rate | Time from the first treatment up to 24 weeks
  Surgical conversion rate, defined as the proportion of patients who achieved gross complete resection after 4-6 cycles of study induction therapy.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | through study completion, an average of 1 year
  Objective response rate (ORR) was defined as complete response (CR) and partial response (PR) proportion of participants.
Disease control rate (DCR) | through study completion, an average of 1 year
  Disease control rate (DCR) was defined as the proportion of patients with complete response (CR), partial response (PR) and stable disease (SD).
R0 surgical conversion rate | Time from the first treatment up to 24 weeks
  R0 surgical conversion rate: defined as the proportion of patients who achieved R0 surgical resection after 4-6 cycles of study induction therapy.
progression free survival(PFS) | From date of the first treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-free survival (PFS), defined as the time from the first initiation of study regimen treatment to the first imaging disease progression or the time of death, whichever occurs first.
Overall Survival (OS) | Survival was followed (every 60±7 days ) up to 24 months after the end of treatment
  Overall survival (OS), defined as the time from the first initiation of the study regimen to death from any cause time.
Adverse Event | through study completion, an average of 1 year
  From the first dose to the end of the study treatment, treatment emergent adverse event（TEAE）、study drug-related adverse event (TRAE) and serious adverse event （SAE) will be summarized and incidence will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Heshui Wu, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol